CLINICAL TRIAL: NCT04858178
Title: Transcutaneous Spinal Neuromodulation to Normalize Autonomic Phenotypes
Brief Title: Transcutaneous Spinal Cord Neuromodulation to Normalize Autonomic Phenotypes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Ryan Solinsky, Clinician-Investigator, Spaulding Rehabilitation Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021P001100
Record Dates: First submitted 2021-04-14; First posted 2021-04-26 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Spinal Cord Injuries; Autonomic Imbalance; Autonomic Dysreflexia; Orthostatic; Hypotension, Neurogenic
MeSH Terms: conditions — Spinal Cord Injuries; Autonomic Dysreflexia; Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Individuals with spinal cord injury (Experimental)
  Interventions: Diagnostic Test: Tests of sympathetic inhibition; Diagnostic Test: Tests of sympathetic activation; Diagnostic Test: Testing of autonomic dysreflexia; Device: Transcutaneous spinal cord stimulation
- Individuals without spinal cord injury (Experimental)
  Interventions: Diagnostic Test: Tests of sympathetic inhibition; Diagnostic Test: Tests of sympathetic activation; Device: Transcutaneous spinal cord stimulation

INTERVENTIONS:
Diagnostic Test: Tests of sympathetic inhibition — Bolus phenylephrine infusion using the Oxford technique will generate the need to inhibit sympathetic activity. Similarly, resting state Mayer waves will be assessed with regard to heart rate and blood pressure responses.
Diagnostic Test: Tests of sympathetic activation — Cold pressor test of the hand will be used to cause sympathetic activation. Valsalva's maneuver will assess the ability to buffer against blood pressure fall (phase II).
Diagnostic Test: Testing of autonomic dysreflexia — Cold pressor test of the foot and bladder pressor response (in individuals with SCI) will be tested.
  Arms: Individuals with spinal cord injury
Device: Transcutaneous spinal cord stimulation — Transcutaneous spinal cord stimulation will be applied at T7-L1 spinal segments to assess alterations in autonomic neuroregulation.

SUMMARY:
This study looks to characterize autonomic nervous system dysfunction after spinal cord injury and identify the potential role that transcutaneous spinal cord stimulation may play at altering neuroregulation. The autonomic nervous system plays key parts in regulation of blood pressure, skin blood flow, and bladder health- all issues that individuals with spinal cord injury typically encounter complications. For both individuals with spinal cord injury and uninjured controls, experiments will utilize multiple parallel recordings to identify how the autonomic nervous system is able to inhibit and activate sympathetic signals. The investigators anticipate that those with autonomic dysfunction after spinal cord injury will exhibit abnormalities in these precise metrics. In both study populations, transcutaneous spinal cord stimulation will be added, testing previously advocated parameters to alter autonomic neuroregulation. In accomplishing this, the investigators hope to give important insights to how the autonomic nervous system works after spinal cord injury and if it's function can be improved utilizing neuromodulation.

ELIGIBILITY:
Inclusion Criteria:

All participants

- age 18-30 years old.

Participants with spinal cord injury

* Adult onset, traumatic spinal cord injury.
* Time since injury 1 year, in an effort to limit baroreflex desensitization.
* American Spinal Injury Association Impairment Scale, A, to limit potential confounders.
* Neurological level of injury, T1-T6, as defined by the International Standards for Neurological Classification of Spinal Cord Injury.

Exclusion Criteria:

* History of cardiovascular disease, hypertension, neurologic disorders (with exception of spinal cord injury), or diabetes.
* Women who are pregnant or lactating.
* Currently taking blood thinners.
* Taking anti-hypertensive or other medication that could influence any of the dependent autonomic variables.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Valsalva Maneuver Phase II | Through study completion, average 3 months
  Presence or absence of phase II on Valsalva maneuver testing, which takes approximately 15 seconds to complete. This will be repeated x3.

SECONDARY OUTCOMES:
Muscle sympathetic nerve activity | Through study completion, average 3 months
  Microneurography will be performed to characterize cardiovascular autonomic phenotypes between uninjured controls and individuals with spinal cord injury. This will be quantified by spike frequency.
Beat-to-beat heart rate | Through study completion, average 3 months
  Electrocardiogram will record continuous measures with changes in R-R interval (ms) quantified and compared to baseline.
Beat-to-beat blood pressure | Through study completion, average 3 months
  Non-invasive continuous blood pressure monitors will be used, with changes in systolic and diastolic pressure (in mmHg) from resting baseline measured.
Continuous galvanic skin response | Through study completion, average 3 months
  Changes from resting state conductance with be quantified with a smartwatch.
Quantify autonomic dysreflexia and orthostatic hypotension | Baseline, prior to initial laboratory diagnostic testing session
  Participants will be given the Autonomic Dysfunction Following Spinal Cord Injury questionnaire (score range 0-436, with higher scores indicating more autonomic dysfunction).
Quantify secondary autonomic complications | Baseline, prior to initial laboratory diagnostic testing session
  Participants will be given the Composite Autonomic Symptom Score (range 0-100, with higher scores indicating more autonomic dysfunction).

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Solinsky, MD, Principal Investigator — Spaulding Rehabilitation Hospital / Harvard Medical School
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No